CLINICAL TRIAL: NCT00912366
Title: A Prospective, Single Center, Observational Study Comparing the Safety and Efficacy of CVATS, HVATS and Open Surgery for Subjects Diagnosed With NSCLC Scheduled to Undergo a Lobectomy
Brief Title: Assessment of Video Assisted Thoracoscopic Surgery (VATS) Versus Open Surgery for Patients Undergoing Lobectomy
Status: Terminated | Type: Observational
Why Stopped: Slow Enrollment
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: AS08015
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: VATS; Lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: VATS
  Interventions: Procedure: Lobectomy
- Group B: Open Surgery
  Interventions: Procedure: Lobectomy

INTERVENTIONS:
Procedure: Lobectomy — Assessment of VATS versus open surgery.
  Other Names: CVATS; HVATS

SUMMARY:
Assessment of VATS versus standard open surgery for treatment of non small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older.
* Subject must have been clinically diagnosed with stage I to stage IIA non small cell lung cancer measuring and judged to be resectable.
* Subject must be able to tolerate general anesthesia, and have cardiopulmonary reserve to tolerate a lobectomy

Exclusion Criteria:

* Subject is pregnant (documented by pregnancy test) or breastfeeding.
* Subject has other severe illnesses that would preclude surgery such as

  * Unstable angina
  * Myocardial Infarction within 3 months
  * Coronary Artery Bypass Graft Surgery
* Subject has other active cancers
* Subject is unable to comply with any of the following:

  * Study requirements
  * Give valid informed consent
  * Follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred for lobectomies at the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Assess hospital length of stay (LOS). | 1 time point (discharge)
Pain Scale Evaluation | 5 time points out to 6 months

SECONDARY OUTCOMES:
Assess quality of life. | 2 time points out to 6 months
Assess peri-operative and post-operative complications. | 5 time points out to 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University School of Medicine, New York, New York, United States